CLINICAL TRIAL: NCT03784196
Title: Whiplash Associated Disorders - Sensory Changes During Rehabilitation
Brief Title: Changes of Pain Sensitivity During Rehabilitation of Patients Suffering From Whiplash Associated Disorders
Status: Completed | Type: Observational
Sponsor: Universidad San Jorge (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: PI16/0132
Record Dates: First submitted 2018-12-10; First posted 2018-12-21 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Whiplash; Whiplash Injury; Neck Pain; Healthy
Keywords: WAD; rehabilitation; whiplash; neck pain; pain sensitivity
MeSH Terms: conditions — Whiplash Injuries; Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Whiplash Associated Disorders: People suffering from acute WAD at the time of recruitment.
  Interventions: Other: Conservative rehabilitation
- Healthy controls: Participants with no neck pain during the past 6 months, chronic pain or other medical disorders relevant to this study.

INTERVENTIONS:
Other: Conservative rehabilitation — WAD participants underwent 2-weeks rehabilitation.
  Groups: Acute Whiplash Associated Disorders

SUMMARY:
This study investigates the sensory profile of people suffering from whiplash associated disorders (WAD) during rehabilitation.

DETAILED DESCRIPTION:
Altered pain sensitivity is commonly reported in WAD populations when compared to a healthy control group but how/if this changes over time during rehabilitation is unclear. This study investigates the effect of 2 weeks rehabilitation protocol on pain sensitivity in a group suffering from WAD compared to a healthy control group.

ELIGIBILITY:
Inclusion Criteria:

WAD

* No more than 3 weeks since MVA/WAD
* WAD grade II defined by Quebec Task Force classification

Controls • Being healthy and free from any pain specific to the low back and/or in general

Exclusion Criteria:

Applies for both groups:

* Pain related to a specific pathology such as spinal stenosis, metastasis, fracture, nerve lesions or injuries to the brain etc.
* Previous painful condition (including neck pain) in the previous 6 months.
* Prior surgery in the neck or shoulder area.
* Radiculopathy.
* Multiple painful sites/areas unrelated to the neck pain.
* Operation to the spine.
* Any neurological or systemic diseases which can affect the outcome measures.
* Pregnancy.
* Lack of ability to cooperate.

Additional exclusion criteria for Controls:

• No current or previous history of on-going pain, defined as pain in the neck/shoulder region and/or elsewhere during the past 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Acute WAD following a motor vehicle accident (MVA) and age- and sex-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Changes in Pressure Pain Thresholds | Baseline, 2 weeks, 6 months
  Changes in pressure pain thresholds will be determined with pressure algometry bilaterally over the neck and leg. PPT is defined as the exact time point where the pressure is first being perceived at painful.
Changes in Conditioned Pain Modulation | Baseline, 2 weeks, 6 months
  Changes in condition pain modulation (CPM) will be measures by recording PPT bilaterally over the neck and leg prior to and following a painful stimuli (a pressure cuff is inflated around the upper arm to create the conditioned stimulus). CPM value is calculated by subtracting raw PPT (without painful stimuli) from PPT under the conditioned stimulus.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Baseline, 2 weeks, 6 months
  A validated and reliable questionnaire that estimates the impact of neck pain on normal daily activities (self-rated disability). NDI consists of 10 dimensions that all are score from 0-5 giving a maximum score of 50. The overall score indicates the level of disability. Below 5 = no disability whereas increased scores indicates increased levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Steffan W Christensen, PhD, Study Director — Aalborg University
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
There are currently no plan on sharing data from this study with other researchers.